CLINICAL TRIAL: NCT03933059
Title: Suicide and Trauma Reduction Initiative Among VEterans
Acronym: STRIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: The Boeing Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 300841
Record Dates: First submitted 2019-04-18; First posted 2019-05-01 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2023-05

CONDITIONS: Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- R&R Park City, Utah (Active Comparator): This group will receive 12 daily individual sessions of CPT at the National Ability Center in Park City, Utah. They will also participate in daily recreational activities.
  Interventions: Other: Psychotherapy
- R&R Salt Lake City, Utah (Active Comparator): This group will receive 12 daily individual sessions of CPT at the National Center for Veterans Studies located on the University of Utah campus in Salt Lake City, Utah.
  Interventions: Other: Psychotherapy
- Weekly Treatment Salt Lake City, Utah (Active Comparator): This group will receive 12 individual sessions of CPT on a weekly basis at the National Center for Veterans Studies located on the University of Utah campus in Salt Lake City, Utah.
  Interventions: Other: Psychotherapy

INTERVENTIONS:
Other: Psychotherapy — Cognitive Processing Therapy is a primarily cognitive form of Cognitive Behavioral Therapy, which has been shown to be effective at reducing symptoms of PTSD.

SUMMARY:
The present study is a pragmatic clinical trial that will examine the effectiveness of Cognitive Processing Therapy (CPT) in reducing PTSD symptom severity, depression symptoms, and suicidal thoughts among military personnel and veterans with PTSD when delivered in three different formats: (1)12 sessions delivered once per week in an office/clinic setting; (2) 12 sessions delivered once per day in an office/clinic setting; and (3) 12 sessions delivered once per day in a recreational setting.

DETAILED DESCRIPTION:
Cognitive behavioral treatments tend to be the most highly efficacious treatments for posttraumatic stress disorder (PTSD). Cognitive Processing Therapy (CPT) is one such treatment that has garnered a significant amount of empirical support, with a recent metaanalysis showing it was among the most effective treatments for PTSD (Watts et al., 2013). Despite its efficacy, many military personnel and veterans with PTSD will not receive CPT (or other recommended treatments) for a variety of reasons. It is possible that adapting CPT from its traditional weekly or biweekly format might both enhance the provision of CPT and reduce barriers to treatment. Specifically, treatment that is compressed into a relatively shorter window may be easier for service members and veterans to complete.

In light of these possibilities, the National Center for Veterans Studies (NCVS) at The University of Utah created the R&R program, an intensive, two-week treatment program for service members and veterans diagnosed with PTSD in partnership with the National Ability Center (NAC), a nonprofit recreational and adaptive sports center located in Park City, Utah. The R&R Program provides CPT in a format designed to circumvent logistical barriers to care and to maximize treatment completion. Preliminary results from 20 service members or veterans who have completed the program show that approximately 70% no longer met criteria for PTSD after completing the program, and suicide ideation decreased significantly (Bryan et al., 2018). Treatment gains during R&R were superior to those found in CPT randomized trials.

The present study seeks to build and broaden current research on CPT. First, it will directly compare the effectiveness of traditional 12-session weekly outpatient CPT against intensive, daily delivery of CPT over 12 days. Second, it will test whether the use of recreational activities improves intensive care by comparing intensive treatment at the NAC with recreational activities against intensive treatment in Salt Lake City without recreational activities. Finally, it will provide important data on the long-term effects of treatment, by assessing PTSD, depression, and suicidal thoughts and behaviors at posttreatment, and 6, 12, and 24 months posttreatment.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older;
2. Current or prior service in the U.S. military;
3. Currently meet criteria for a diagnosis of posttraumatic stress disorder (as determined by the CAPS-5);
4. Be able to complete the informed consent process.

Exclusion Criteria:

1. Current substance dependence disorder;
2. Severe suicide ideation during the past two weeks (as determined by the BSSI and clinical interview) warranting hospitalization;
3. Suicide attempt during the previous three months;
4. Impaired mental status that precludes ability to provide informed consent (e.g., intoxication, psychosis, mania).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in PTSD symptom severity since baseline measured by the Clinician Administered PTSD Scale | Past month symptoms, assessed within a month of completing treatment, and 6-months, 12-months, 18-months, and 24 months after completing treatment
  Interviewer administered measure to determine the severity of PTSD. Items are summed to create a total score (Range: 0-80) where higher scores indicate greater symptom severity.
Change in PTSD symptom severity since baseline measured by the Clinician Administered PTSD Scale | Past week symptoms, assessed the last day of treatment for those completing the two week treatment retreats
  Interviewer administered measure to determine the severity of PTSD. Items are summed to create a total score (Range: 0-80) where higher scores indicate greater symptom severity.

SECONDARY OUTCOMES:
Change in suicidal thoughts and behaviors since baseline measured by the Scale for Suicidal Ideation | Past week symptoms, assessed within a month of completing treatment, and 6-months, 12-months, 18-months, and 24 months after completing treatment
  Self-report assessment of severity of suicidal thoughts and behaviors. Items are summed (range: 0-63) and higher scores indicate greater suicide severity.
Change in depression symptom severity since baseline measured by the Patient Health Questionnaire | Past two week symptoms, assessed within a month of completing treatment, and 6-months, 12-months, 18-months, and 24 months after completing treatment
  Self-report assessment of depression symptom severity. Items are summed (range: 0-27) and higher scores indicate greater depression symptom severity.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Bryan CJ, Leifker FR, Rozek DC, Bryan AO, Reynolds ML, Oakey DN, Roberge E. Examining the effectiveness of an intensive, 2-week treatment program for military personnel and veterans with PTSD: Results of a pilot, open-label, prospective cohort trial. J Clin Psychol. 2018 Dec;74(12):2070-2081. doi: 10.1002/jclp.22651. Epub 2018 Jun 19. PMID 29917224